CLINICAL TRIAL: NCT03520361
Title: Comparative Evaluation of the Efficacy of Oral Sulfate Solution (OSS) and 2L Polyethylene Glycol (PEG) With Ascorbic Acid (Asc) for Bowel Preparation of Elderly People: A Multicenter Prospective Randomized Study
Brief Title: Comparison Between OSS and 2L PEG/Asc for Bowel Preparation of Elderly People
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: KangWon National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017-03-011
Record Dates: First submitted 2017-08-20; First posted 2018-05-09 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Bowel preparation; Oral sulfate solution; Polyethylene glycol; Ascorbic acid

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single Blind (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral sulfate solution (OSS) taking group (Experimental): On the evening before colonoscopy, drink 177ml of OSS (Suclear®) (473ml including water in container), additionally allow another 946 ml of water. On the day of colonoscopy, drink 177ml of OSS (473ml including water in container), additionally allow another 946 ml of water.
  Interventions: Drug: Oral sulfate solution (OSS)
- 2L PEG/Asc taking group (Active Comparator): On the evening before colonoscopy, drink 1L of 2L PEG/Asc (Haprep®) solution, additionally allow another 500 ml of water. On the day of colonoscopy, drink 1L of 2L PEG/Asc solution, additionally allow another 500 ml of water.
  Interventions: Drug: 2L PEG/Asc

INTERVENTIONS:
Drug: Oral sulfate solution (OSS) — Compositions/177ml : Sodium sulfate 17.5g, Potassium sulfate 3.13g, Magnesium sulfate 1.6g
  Other Names: Suclear® solution (Phambio Korea, Seoul, Korea)
  Arms: Oral sulfate solution (OSS) taking group
Drug: 2L PEG/Asc — Compositions/1L : Sodium chloride 2.89g, Potassium chloride 1.015g, Anhydrous sodium sulfate 7.5g, Polyethylene glycol 3350 100g, Ascorbic acid 4.7g, Sodium ascorbate 5.9g
  Other Names: Haprep® powder (Phambio Korea, Seoul, Korea)
  Arms: 2L PEG/Asc taking group

SUMMARY:
For evaluation of the usefulness of oral sulfate solution (OSS) for bowel preparation of elderly people, investigators compare the efficacy, tolerability and safety between OSS and 2L polyethylene glycol (PEG) with ascorbic acid (Asc).

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized parallel arm, investigator initiated trial.

The aim of study is to compare oral sulfate solution (OSS) with 2L polyethylene glycol (PEG) with ascorbic acid (Asc) for bowel preparation in elderly people.

99 participants will be enrolled in each group (198 in total). The primary outcome is the efficacy of bowel preparation. Secondary outcomes are tolerability, satisfaction, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy examinee aged 65-80
* Examinee agree with informed consent

Exclusion Criteria:

* Cognitive disorder, mental retardation
* Bowel obstruction
* Severe constipation (<3 bowel movements per week with or without regular or intermittent laxatives)
* History of bowel surgery
* Liver cirrhosis or ascites
* Heart failure, cardiac disease (ischemic heart disease or coronary artery disease within the last 6 months)
* Inflammatory bowel disease
* Pregnancy, lactating woman
* Renal impairment or history of impaired renal function
* History of hypersensitivity reaction to bowel preparation

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation scale of right/transverse/left colon using Boston bowel preparation scale (BPPS) | 3 months
  The BBPS assesses cleanliness of 3 segments of the colon (ascending, transverse, and descending colon), and the total is a 10-point scale (0-9) that grades each segment of the colon from 0 to 3. In this study, adequate bowel preparation is defined as a total score 6 points or higher and individual score of 2 points or higher in each segment.

SECONDARY OUTCOMES:
Subject's satisfaction based on the 10-point visual analog scale | 3 months
  The 10-point scale from 0 to 10
Number of subjects who have a difficulty taking solution based on the 5-grade scale | 3 months
  The 5-grade scale: very easy, easy, moderate, hard, and very hard
Taste of recommended bowel preparation agent based on the 5-grade scale | 3 months
  The 5-grade scale: very good, good, neutral, bad, and very bad
Number of subjects who have a willingness to repeat the same regimen | 3 months
  using questionnaires: yes, no
Rate of subjects with nausea | 3 months
  using questionnaires: yes, no
Rate of subjects with vomiting | 3 months
  using questionnaires: yes, no
Rate of subjects with abdominal pain | 3 months
  using questionnaires: yes, no
Rate of subjects with abdominal distention | 3 months
  using questionnaires: yes, no
Rate of subjects with thirst | 3 months
  using questionnaires: yes, no
Rate of subjects with dizziness | 3 months
  using questionnaires: yes, no
Rate of subjects with paresthesia | 3 months
  using questionnaires: yes, no
Sodium level in mmol/L | an average of 1 year
  change in electrolyte values before and after bowel preparation
Potassium level in mmol/L | 3 months
  change in electrolyte values before and after bowel preparation
Chloride level in mmol/L | 3 months
  change in electrolyte values before and after bowel preparation
Magnesium level in mg/dL | 3 months
  change in electrolyte values before and after bowel preparation
Phosphorus level in mg/dL | 3 months
  change in electrolyte values before and after bowel preparation
Calcium level in mg/dL | 3 months
  change in electrolyte values before and after bowel preparation
Blood urea nitrogen level in mg/dL | 3 months
  change in electrolyte values before and after bowel preparation
Creatinine level in mg/dL | 3 months
  change in electrolyte values before and after bowel preparation
Serum osmolarity in mmol/kg | 3 months
  change in osmolarity values before and after bowel preparation
Urine osmolarity in mmol/L | 3 months
  change in osmolarity values before and after bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Sung Chul Park, MD, PhD, Principal Investigator — KangWon National University Hospital
Locations (1):
- Kangwon National University Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided